CLINICAL TRIAL: NCT01016535
Title: Care of Child's Hygiene From Zero to Two Years Old: Health Professionals' Perceptions of the Strategy and the Family Caregivers
Brief Title: Care of Child's Hygiene From Zero to Two Years Old
Acronym: CCH
Status: Completed | Type: Observational
Sponsor: Faculdade Santa Marcelina (Other)
Responsible Party: GIANA MARROCHI, FACULDADE SANTA MARCELINA
Other Study IDs: FASM1
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Children Health Under Two Years Old; Health Professionals
Keywords: Family Health Program; Hygiene; Child Health

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Children, Health Professionals

SUMMARY:
This study aimed to identify the perceptions of family caregivers and professionals of the Family Health Strategy (FHS) for health care for children from 0 to 2 years, and actions on this issue developed by the FHS.

DETAILED DESCRIPTION:
This study aimed to identify the perceptions of family caregivers and professionals of the Family Health Strategy (FHS) for health care for children from 0 to 2 years, and actions on this issue developed by the FHS. Chosen by a descriptive exploratory with a qualitative approach, consisting of 19 subjects while they were 9 professionals and 10 family caregivers. For data collection was used a semi-tour interview and for the treatment of empirical data, the technique of content analysis recommended by Bardin. For presentation and discussion of results the categories from the speech made the interviewers grouped as the possibility of confrontation between the speaches of the two groups, total of 6 categories: hygienist model: focus on personal hygiene, model medicocêntrico x extended care, environmental risk: the care with hygiene and socioeconomic conditions, family and life experience influence care with hygiene, process work x on caregiver perception of guidance received by the health service, link child / caregiver. The perceptions found in the discourse of professionals and caregivers showed that the biologically vision and focus on the body prevalent in health care, and that such care is still centered in the figure of the doctor because of the historical and cultural hegemony curative.

ELIGIBILITY:
Inclusion Criteria:

* children under two years old
* professional member of the healthcare team

Exclusion Criteria:

* caregivers who were not relatives
* children who had any physical impairment and/or mental

Ages: 1 Month to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children's caregivers from zero to two years old monitored in a health center health professionals of a team of a health center
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GIANA MARROCHI, Principal Investigator — Faculdade Santa Marcelina
Locations (1):
- Faculdade Santa Marcelina, São Paulo, São Paulo, Brazil